CLINICAL TRIAL: NCT00530647
Title: fMRI Study of Brain Neural Network and Plasticity After Stroke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Other Study IDs: 2006-08-133
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Last update posted 2007-09-17 (Estimated); Status verified 2006-10

CONDITIONS: Stroke
Keywords: Brain motor network, Plasticity, functional MRI, Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purposes of this study are to investigate the functional connectivity of motor network in patients of stroke and investigate the mechanism of brain plasticity for recovery after stroke.

ELIGIBILITY:
Inclusion Criteria:

* 1st-ever-stroke
* whose corticospinal tract was injured
* less than 1 month after stroke onset

Exclusion Criteria:

* Claustrophobia
* who use cardiac pacemaker
* intracranial metal
* uncontrolled hypertension or hypotension

Ages: 20 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Suk Hoon Ohn, MD, MS, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Seoul, South Korea